CLINICAL TRIAL: NCT02414841
Title: Multicenter, Double Blind, Placebo Controlled Study of Vonapanitase (PRT- 201) Administered Immediately After Radiocephalic Arteriovenous Fistula Creation in Patients With Chronic Kidney Disease
Brief Title: A Study of Vonapanitase (PRT-201) Administered Immediately After Radiocephalic Arteriovenous Fistula(AVF) Creation in Patients With Chronic Kidney Disease (CKD) (PATENCY-2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Proteon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRT-201-320
Record Dates: First submitted 2015-04-08; First posted 2015-04-13 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Chronic Kidney Disease
Keywords: radiocephalic; arteriovenous fistula; AVF; hemodialysis; PRT-201; vonapanitase; vascular access; kidney; renal; PATENCY-2; secondary patency; fistula abandonment; use for hemodialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Arteriovenous Fistula | interventions — cholesterol-binding protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vonapanitase (Active Comparator): Vonapanitase administered at the time of radiocephalic fistula creation
  Interventions: Drug: Vonapanitase
- Placebo (Placebo Comparator): Placebo administered at the time of radiocephalic fistula creation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vonapanitase
  Other Names: PRT-201
  Arms: Vonapanitase
Drug: Placebo
  Arms: Placebo

SUMMARY:
This research study is designed to assess the safety and effectiveness of an experimental drug called vonapanitase (PRT-201) in patients both receiving or expecting to receive hemodialysis who have chronic kidney disease and who are undergoing surgery to create a new access point to their bloodstream for hemodialysis. Vonapanitase is a protein that has been shown in previous research studies to help keep vessels patent when applied to the outside surface of the blood vessels (arteries and veins) in patients who undergo surgery to create an arteriovenous fistula (AVF). The purpose of this study is to determine whether vonapanitase when applied to a limited segment of your blood vessel (about 2 inches) immediately after surgery is safe and improves the patency of your AVF.

ELIGIBILITY:
Inclusion Criteria:

1. Age of at least 18 years.
2. Life expectancy of at least 6 months.
3. Diagnosis of CKD.
4. Planned creation of a new radiocephalic AVF (revision of an existing AVF is not eligible).
5. Ability to understand and comply with the requirements of the entire study and to communicate with the study team.
6. Written informed consent using a document that has been approved by the Institutional Review Board (IRB) or Independent Ethics Committee (IEC).
7. If female and of childbearing potential (premenopausal and not surgically sterile) must have a negative serum pregnancy test at the screening visit and be willing to use contraception from the time of the screening visit to 2 weeks following study drug administration. Acceptable methods of birth control include abstinence, barrier methods, hormones, or intra-uterine device.

Exclusion Criteria:

1. Malignancy or treatment for malignancy within the previous 12 months with the exception of the following cancers if they have been resected: localized basal cell or squamous cell skin cancer, or any cancer in situ.
2. Presence of any significant medical condition that might significantly confound the collection of safety and efficacy data in this study.
3. Previous treatment with vonapanitase (PRT-201).
4. Treatment with any investigational drug within the previous 30 days or investigational antibody therapy within the previous 90 days prior to signing informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 696 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2019-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (36):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - AKDHC Medical Research Services, LLC, Phoenix, Arizona
  - Banner University Medical Center Tucson, Tucson, Arizona
  - AKDHC Medical Research Services, LLc, Tucson, Arizona
  - VA Loma Linda Healthcare System, Loma Linda, California
  - VA Medical Center Long Beach, Long Beach, California
  - Keck University Hospital at USC, Los Angeles, California
  - Kaiser Permanente, San Diego, California
  - California Institute of Renal Research, San Diego, California
  - Kaiser Permanente Northern California, San Francisco, California
  - University of Chicago, Chicago, Illinois
  - RenalCare Associates, S.C., Peoria, Illinois
  - Lutheran Hospital Network of Indiana, Fort Wayne, Indiana
  - The University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Louisville, Louisville, Kentucky
  - Tulane University, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Greenwood Leflore Hospital, Greenwood, Mississippi
  - Saint Luke's Hospital, Kansas City, Missouri
  - New York Presbyterian Hospital-Weill Cornell Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - VA Pittsburg Healthcare System, Pittsburgh, Pennsylvania
  - SC Nephrology and Hypertension Center, Inc., Orangeburg, South Carolina
  - Knoxville Kidney Center, Knoxville, Tennessee
  - Cardiothoracis and Vascular Surgeons, Austin, Texas
  - Baylor College of Medicine, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - Lake Washington Vascular Center, Bellevue, Washington
  - University of Wisconsin School of Medicine and PH, Madison, Wisconsin
- Canada (5):
  - University of Alberta, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - London Health Science Center, London, Ontario
  - University Health Network Toronto General Hospital, Toronto, Ontario
  - McGill University Health Centre- Royal Victoria Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Heindel P, Fitzgibbon JJ, Secemsky EA, Belkin M, Ozaki CK, Hussain MA. Evaluating the effectiveness of systemic heparin during arteriovenous fistula creation by emulating a target trial. Am J Epidemiol. 2025 Mar 4;194(3):651-658. doi: 10.1093/aje/kwae098. PMID 38825327
- [Derived] Heindel P, Fitzgibbon JJ, Feliz JD, Hentschel DM, Burke SK, Al-Omran M, Bhatt DL, Belkin M, Ozaki CK, Hussain MA. Evaluating national guideline concordance of recurrent interventions after radiocephalic arteriovenous fistula creation. J Vasc Surg. 2023 Apr;77(4):1206-1215.e2. doi: 10.1016/j.jvs.2022.12.017. Epub 2022 Dec 22. PMID 36567000
- [Derived] Peden EK, Lucas JF 3rd, Browne BJ, Settle SM, Scavo VA, Bleyer AJ, Ozaki CK, Teruya TH, Wilson SE, Mishler RE, Ferris BL, Hendon KS, Moist L, Dixon BS, Wong MD, Magill M, Lindow F, Gustafson P, Burke SK; PATENCY-2 Investigators. PATENCY-2 trial of vonapanitase to promote radiocephalic fistula use for hemodialysis and secondary patency. J Vasc Access. 2022 Mar;23(2):265-274. doi: 10.1177/1129729820985626. Epub 2021 Jan 22. PMID 33482699

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 696 patients signed informed consent; 613 patients were randomized; 603 were treated
Pre-assignment Details: Participants were excluded if they did not have a radiocephalic fistula created at the time of surgery
Groups:
- Vonapanitase: Vonapanitase administered at the time of radiocephalic fistula creation
  vonapanitase
- Placebo: Placebo administered at the time of radiocephalic fistula creation
  Placebo
Period: Overall Study
Arm/Group | Vonapanitase | Placebo
Started | 405 | 208
Completed | 349 | 175
Not Completed | 56 | 33
Not completed — Withdrawal by Subject | 7 | 5
Not completed — Lost to Follow-up | 13 | 6
Not completed — Death | 17 | 14
Not completed — Received a Kidney Transplant | 13 | 4
Not completed — Randomized But Not Treated | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vonapanitase | Placebo | Total
Number analyzed (Participants) | 405 | 208 | 613
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 277 | 132 | 409
  >=65 years | 128 | 76 | 204
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 46 | 147
  Male | 304 | 162 | 466
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 19 | 10 | 29
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 104 | 45 | 149
  White | 269 | 149 | 418
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 3 | 10
Region of Enrollment [Number; unit: participants]
  Canada | 41 | 18 | 59
  United States | 358 | 186 | 544

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimate of Secondary AVF Patency
Description: Kaplan-Meier estimate of median time from AVF creation until AVF abandonment (secondary patency)
Time Frame: Median time from AVF creation to AVF abandonment (secondary patency), assessed up to 1 year.
Population: Full analysis set includes all 613 patients who were randomized
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Placebo: Placebo administered at the time of radiocephalic fistula creation. The placebo is identical in appearance and composition of vonapanitase but lacks the active ingredient.
  Placebo
Arm/Group | Vonapanitase | Placebo
Number analyzed (Participants) | 405 | 208
Days | NA [NA to NA] — The median time to the event based on Kaplan-Meier estimates was not reached in this trial | NA [NA to NA] — The median time to the event based on Kaplan-Meier estimates was not reached in this trial
Statistical Analysis 1: Comparison: Vonapanitase vs Placebo; Test type: Superiority; p = 0.932, Log Rank; Weighted; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.67 to 1.39] — Performed as sensitivity analysis

2. Primary Outcome: Number of Participants With AVF Use for Hemodialysis
Description: AVF use for hemodialysis is defined as the ability of the study AVF to be successfully cannulated and used for hemodialysis for a minimum of 90 days or at least 30 days prior to a patient's last visit, if hemodialysis has not been initiated at least 90 days prior to the patient's last visit. If AVF use is not defined as above, non-use of the AVF for hemodialysis is defined as an abandoned fistula prior to use; or if hemodialysis is recorded on 2 consecutive visits and there is no cannulation date or duration of use is less than 90 days. The patients who are not categorized as having use or non-use of the AVF have insufficient data to determine AVF use for hemodialysis and will be categorized as having indeterminate use.
Time Frame: Assessed at up to 12 Months
Population: Patients having use or non-use of their AVF. Patients with indeterminate use of their AVF were excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Vonapanitase | Placebo
Number analyzed (Participants) | 405 | 208
Participants
  AVF Used | 209 | 99
  AVF Not Used | 91 | 53
  Indeterminant AVF Use | 105 | 56
Statistical Analysis 1: Comparison: Vonapanitase vs Placebo; Test type: Superiority; p = 0.328, Chi-squared

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) through Week 4; Only AEs associated with the AVF extremity Week 4-Month 12.
Groups:
- Placebo: Placebo administered at the time of radiocephalic fistula creation. The placebo is identical in appearance and composition of vonapanitase but lacks the active ingredient.
Arm/Group | Vonapanitase | Placebo
All-Cause Mortality (participants affected / at risk) | 17/399 | 14/204
Serious Adverse Events (participants affected / at risk) | 48/399 | 30/204
Other Adverse Events (participants affected / at risk) | 247/399 | 135/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vonapanitase (N=399) | Placebo (N=204)
Pulseless Electrical Activity (Cardiac disorders) | 0 | 1
Fluid Overload (Metabolism and nutrition disorders) | 0 | 3
Sepsis (Infections and infestations) | 2 | 1
Cardiac Arrest (Cardiac disorders) | 2 | 5
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Renal Failure (Renal and urinary disorders) | 1 | 2
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Venous Thrombosis (Vascular disorders) | 0 | 1
Steal Syndrome (Vascular disorders) | 1 | 1
Toe Surgery (Surgical and medical procedures) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 4 | 4
Cerebral Haemorrhage (Nervous system disorders) | 0 | 1
Renal Failure Chronic (Renal and urinary disorders) | 1 | 2
Arteriovenous Fistula Thrombosis (Injury, poisoning and procedural complications) | 7 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Pulmonary Tuberculosis (Infections and infestations) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 1 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Septic Shock (Infections and infestations) | 0 | 1
Haematoma (Vascular disorders) | 0 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Calciphylaxis (Metabolism and nutrition disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Device Kink (General disorders) | 1 | 0
Collateral Circulation (Vascular disorders) | 2 | 0
Confusional State (Psychiatric disorders) | 1 | 0
Vascular Stenosis (Vascular disorders) | 2 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 2 | 0
Syncope (Nervous system disorders) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Chest Pain (General disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Unknown Cause of Death (General disorders) | 1 | 0
Post Procedural Infection (Infections and infestations) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Sudden Death (General disorders) | 1 | 0
Circulatory Collapse (Vascular disorders) | 1 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Azotaemia (Renal and urinary disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Generalised Oedema (General disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vonapanitase (N=399) | Placebo (N=204)
Local Swelling (General disorders) | 20 | 4
Arteriovenous Fistula Thrombosis (Injury, poisoning and procedural complications) | 67 | 38
Vascular Stenosis (Vascular disorders) | 140 | 85
Haematoma (Vascular disorders) | 20 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/41/NCT02414841/Prot_SAP_000.pdf